CLINICAL TRIAL: NCT04117009
Title: Effects of Remifentanil on Diastolic and Systolic Function in Patients With Diastolic Dysfunction
Brief Title: Effects of Remifentanil on Cardiac Function in Patients With Diastolic Dysfunction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Özge Köner, Clinical Professor, Yeditepe University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17AKD137
Record Dates: First submitted 2019-10-02; First posted 2019-10-07 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Diastolic Dysfunction
Keywords: diastolic dysfunction; remifentanil
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Intervention Model Description: Baseline echocardiographic examination will be performed to evaluate the systolic and diastolic function of the left ventricle in the spontaneously breathing subjects right before anesthesia and study drug infusion begins. Then the same participants will be given remifentanil (ultiva at a concentration of 20 micg/ml) at a rate to reach a target plasma level of 2 ng/mL by means of a target controlled Infusion pump. Once the target drug concentration is reached (which is expected to take around 10-15 minutes), the final echocardiographic examination will be performed to assess systolic and diastolic function again.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remifentanil 2 ng/mL (Experimental): Following baseline echocardiographic evaluation, Remifentanil (ultiva at a concentration of 20 micg/ml) infusion will be started at a rate to reach a target plasma level of 2 ng/mL. A target Controlled Infusion pump will be used to infuse the study drug. Once the target drug concentration is reached (which is expected to reach around 10-15 minutes), the final echocardiographic examination will be performed.
  Interventions: Drug: Remifentanil 2 MG; Diagnostic Test: Echocardiographic evaluation
- Baseline (Experimental): Baseline transthoracic echocardiographic examination will be performed in the spontaneously breathing patients right before the surgical procedure and study drug infusion begins.
  Interventions: Diagnostic Test: Echocardiographic evaluation

INTERVENTIONS:
Drug: Remifentanil 2 MG — Once the participants transferred to operating room, electrocardiography, noninvasive blood pressure, pulse oximetry, and respiratory rate will be recorded. An increase or decrease from the baseline value of 30% in mean arterial pressure will be treated with iv boluses of (5 mg) ephedrine or glyceryl trinitrate (25 micg). All the participants will undergo a baseline transthoracic echocardiographic evaluation to assess the systolic and diastolic function of the left ventricle before the infusion of the study drug. Then the patients will be given oxygen by a face mask at a rate of 5-6 L/min, and Remifentanil infusion will be started using a target controlled infusion pump to reach a target plasma concentration of 2 ng/mL. Once the target concentration is reached, second echocardiographic evaluation to assess the systolic and diastolic function will be performed. Potential side effects of Remifentanil will be monitored.
  Other Names: Ultiva 2 mg.; Rentanil 2 mg.; Opiva 2 mg.
  Arms: Remifentanil 2 ng/mL
Diagnostic Test: Echocardiographic evaluation — Transthoracic echocardiographic examination will be performed in the spontaneously breathing patients right before the surgical procedure.

SUMMARY:
In this study ASA 1, 2 individuals with grade 1 or 2 diastolic dysfunction will be recruited to assess the effects of Remifentanil infusion on left ventricular function evaluated with transthoracic echocardiagraphy.

DETAILED DESCRIPTION:
Our aim in this study is to evaluate the effects of Remifentanil infusion on left ventricular function evaluated with transthoracic echocardiagraphy on ASA 1, 2 individuals with grade 1 or 2 diastolic dysfunction. Methods: 30 ASA 1-2 individuals with grade 1 or 2 diastolic dysfunction whose left ventricular ejection fraction is above 50% will be recruited. The patients will be selected among the ones who planned to undergo elective surgery either under general or regional anesthesia.

Patients with atrial fibrillation, atrioventricular block, severe heart valve disease, tachyarrhythmia-bradyarrhythmia, left ventricular ejection fraction < 50% and regional contraction anomaly, patients with liver, renal dysfunction, patients with lung disease, acute coronary syndrome, body mass index >30 kg/m2, no oral intake for solid food more than 8 hours will be excluded from the study.

Baseline echocardiographic examination will be performed in the spontaneously breathing subjects right before the surgical procedure and study drug begins. Then remifentanil infusion will be started at a rate to reach target plasma level of 2 ng/mL. A target Controlled Infusion pump will be used to infuse the study drug. Once the target drug concentration is reached, the final echocardiographic examination will be performed.

After recording the baseline heart rate, respiratory rate, noninvasive blood pressure, pulse oximeter, sedation level, the same parameters will be recorded every 5 minutes during the remifentanil infusion period. Once the final echocardiographic evaluation is performed abovementioned parameters will be recorded for the last time.

Statistical analysis: The sample size calculation is made according to an increase or decrease in E/e' (alpha <0,05; beta= 0,8).

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older ASA 1, 2 adults with first or second degree diastolic dysfunction.

Exclusion Criteria:

* Atrial fibrillation, Atrioventricular block, tachyarrhythmia, bradyarrhythmia, Left ventricular ejection fraction lower than 50%, body mass index >30 kg/m2, Liver, kidney and lung disease.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
A change in diastolic function from the baseline value. | Following baseline measurement, the second measurement will be performed as soon as the 2 ng/mL target plasma level of remifentanil is reached. This will probably take 15 to 20 minutes for each patient until the end of the 6 month long study period.]
  A change from the baseline diastolic function evaluated with echocardiography which is measured as soon as the patient arrives at the operating room when compared to diastolic function measured after reaching the target (2ng/mL) plasma concentration of remifentanil.

SECONDARY OUTCOMES:
A change in systolic function from the baseline value. | Following baseline measurement, the second measurement will be performed as soon as the 2 ng/mL target plasma level of remifentanil is reached. This will probably take 10 to 15 minutes for each patient until the end of the 6 month long study period.
  A change from the baseline systolic function evaluated with echocardiography which is measured as soon as the patient arrives at the operating room when compared to systolic function measured after reaching the target (2ng/mL) plasma concentration of remifentanil.

CONTACTS AND LOCATIONS:
Overall Officials: Özge Köner, Professor, Study Director — Yeditepe University
Locations (1):
- Yeditepe University Hospital, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bolliger D, Seeberger MD, Kasper J, Skarvan K, Seeberger E, Lurati Buse G, Buser P, Filipovic M. Remifentanil does not impair left ventricular systolic and diastolic function in young healthy patients. Br J Anaesth. 2011 Apr;106(4):573-9. doi: 10.1093/bja/aeq414. Epub 2011 Jan 27. PMID 21273230
- [Result] Couture P, Denault AY, Shi Y, Deschamps A, Cossette M, Pellerin M, Tardif JC. Effects of anesthetic induction in patients with diastolic dysfunction. Can J Anaesth. 2009 May;56(5):357-65. doi: 10.1007/s12630-009-9068-z. Epub 2009 Apr 2. PMID 19340494